CLINICAL TRIAL: NCT06211049
Title: Efficacy of Vitex Agnus-castus BNO 1095 (20 mg) in Women With Primary Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bionorica SE (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AgnoMed; 2023-503688-41-00 (Other: European Union and European Economic Area via CTIS); U1111-1288-9484 (Registry Identifier: World Health Organization [WHO] Registry Network)
Record Dates: First submitted 2023-11-23; First posted 2024-01-18 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Primary Dysmenorrhea
Keywords: Vitex agnus-castus; Menstrual pain
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, multicenter, placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitex agnus-castus BNO 1095 (20 mg) (Experimental): 1 tablet once daily for about 4 menstrual cycles (cramping windows of Cycles 3-6) (i.e., 113 days in case of a 28-day menstrual cycle).
  Interventions: Drug: Vitex agnus-castus BNO 1095 (20 mg)
- Placebo (Placebo Comparator): 1 tablet once daily for about 4 menstrual cycles (cramping windows of Cycles 3-6) (i.e., 113 days in case of a 28-day menstrual cycle).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitex agnus-castus BNO 1095 (20 mg) — 1 tablet once daily for about 4 menstrual cycles (cramping windows of Cycles 3-6) (i.e.,113 days in case of a 28-day menstrual cycle).
  Arms: Vitex agnus-castus BNO 1095 (20 mg)
Drug: Placebo — 1 tablet once daily for about 4 menstrual cycles (cramping windows of Cycles 3-6) (i.e.,113 days in case of a 28-day menstrual cycle).
  Arms: Placebo

SUMMARY:
In this Phase III study, the herbal product Vitex agnus-castus BNO 1095 20 mg will be tested.

The sponsor would like to find out if treatment with Vitex agnus-castus BNO 1095 20 mg may improve the cramping pain before or during menstruation (primary dysmenorrhea) (without an organic cause) in women and if this treatment is safe. It is tested, if the pelvic pain and other symptoms during menstruation improve in patients who are treated with Vitex agnus-castus BNO 1095 20 mg and if therefore the standard treatments for primary dysmenorrhea, for example pain relief medications will not have to be increased.

The study has 2 treatment groups. Patients in one group will receive Vitex agnus-castus BNO 1095 20 mg, and patients in the other group will receive a placebo. Placebo tablets look like Vitex agnus-castus BNO 1095 20 mg tablets but have no active ingredient. Patients will be randomly assigned (like tossing a coin) to one of the 2 groups (this process is called randomization). The chance for the patients to receive Vitex agnus-castus BNO 1095 is 50%. Neither the patients nor the investigators know which product the patients are taking (this method is known as "double-blind").

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, multicenter, phase III clinical trial to investigate the efficacy and safety of investigational medicinal product (IMP) Vitex agnus-castus BNO 1095 20 mg in women with primary dysmenorrhea.

The clinical trial will be conducted in Austria, Czech Republic, Germany, Hungary, Poland and Sweden.

About 390 patients will be screened so that about 300 patients (150 patients per treatment group) will be randomized.

Vitex agnus-castus BNO 1095 20 mg is extracted from the fruits of the plant Vitex agnus-castus also called monk's pepper or chaste tree. Vitex agnus-castus BNO 1095 20 mg is currently marketed for the treatment of the premenstrual syndrome (PMS) which means repeated occurrence of physical, behavioral and psychological symptoms the days before the onset of menstruation, but it is not authorized for the treatment of primary dysmenorrhea.

The study has 2 treatment groups. Patients in one group will receive Vitex agnus-castus BNO 1095 20 mg, and patients in the other group will receive a placebo. Patients will be randomly assigned 1:1 to one of the 2 groups. The chance to receive Vitex agnus-castus BNO 1095 is 50%. The study is double blinded, neither the patients nor the investigators know which product the patients are taking.

The study will last about 7 months for each patient. There will be 5 visits at the study site, and in addition the patients will receive 3 phone calls from the study site. On average, each study site visit will take about 2 hours and each phone call about half an hour.

The trial will include 3 phases: a screening and run-in phase of up to 2 menstrual cycles, a treatment phase of 4 menstrual cycles and a follow-up phase of 1 menstrual cycle. The length of each phase depends on the length of women's menstrual cycle. If their menstrual cycle is 28 days, the screening and run-in phase will take up to 59 days (slightly more than 2 menstrual cycles), the treatment phase 113 days (about 4 menstrual cycles), and the follow-up phase 28 days (1 menstrual cycle).

The main objective of this study is to determine if primary dysmenorrhea improves in women treated with Vitex agnus-castus BNO 1095 20 mg compared to placebo over a treatment duration of 3 menstrual cycles (cramping windows of Cycles 3-5).

Vitex agnus-castus BNO 1095 20 mg or placebo tablets are taken orally (means by mouth) once a day during the treatment phase.

If a patient usually takes pain relief medication for primary dysmenorrhea, the patient is allowed to continue taking this pain relief medication during study participation.

The patients will complete the dysmenorrhea daily diary (DysDD) every day in the evening. Depending on her bleeding status, the diary includes questions about menstrual bleeding, pieces of sanitary protection used, severity of the worst pain or cramps in the pelvic area on a numerical rating scale (NRS), intake of pain relief medication, and impact on daily life in an electronic diary (handheld device).

Additionally, the dysmenorrhea associated symptoms nausea, vomiting, diarrhea, fatigue, weakness, fainting, and headache will be assessed by the patients on a NRS in the electronic diary on Days 1-3 of the menstrual cycle. Migraine will be assessed by the investigator at the clinical trial visits. The patient and investigator will assess the efficacy of treatment on a 5-point verbal rating scale at the end of treatment and at the end of the study (EoS).

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-49 years who have the capacity for consenting
2. Patient has been informed of the nature, scope, and relevance of the clinical trial, voluntary agrees in participation and the trial provisions, and has duly signed the approved informed consent form (ICF)
3. Diagnosed primary dysmenorrhea
4. If patients take pain relief medication for primary dysmenorrhea, this medication should be taken unchanged with regard to application form and kind of medication including strength during the Screening as well as during the first three treatment cycles.

   Note: Medication (drugs) for primary dysmenorrhea as mono- or combination therapy in form of tablets/capsules regularly used by the patient before Screening is allowed to be used as standard pain relief medication during the trial apart from non-medication methods. A complete list of allowed pain relief medication is attached to the protocol.

   This medication should be taken by the patient at least for 1 cycle before Screening guaranteeing a stable intake of this medication in total for 3 cycles before randomization.
5. Patients with a regular menstrual cycle duration of ≥24 to ≤38 days
6. Patients agreeing to use one of the following contraception methods throughout the trial:

   1. Bilateral tubal occlusion
   2. Vasectomized partner (provided that the partner is the sole sexual partner of the woman and has received medical assessment of the surgical success)
   3. Sexual abstinence Abstinence is only accepted as true abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods and withdrawal) is not an acceptable method of contraception
   4. Male or female condom with or without spermicide
   5. Cap, diaphragm, or sponge with spermicide

Exclusion Criteria:

A patient will not be eligible for inclusion if any of the following criteria applies:

1. Non-menstruating women
2. Clinically diagnosed secondary dysmenorrhea (e.g., fibroids, uterine adenomyosis, endometriosis, pelvic inflammation, ovarian pathologies, or other pelvic diseases)
3. Dysmenorrhea resulting from the use of an intrauterine device
4. Use of hormonal contraceptives (oral, intravaginal, transdermal, injectable, implantable), intrauterine device, or intrauterine hormone-releasing system within 6 months prior to the trial and not willing to waive it during the entire trial period
5. Any surgical treatments in the past (e.g., due to myoma) that may cause pain, adhesions or scarring in the lower abdomen Note: Further diagnostic examination (e.g., laparoscopy for differential diagnosis, exclusion of endometriosis) if deemed necessary by the investigator will be outside the trial protocol and reimbursement
6. Known or suspected gastrointestinal or urological conditions that may cause abdominal and/or pelvic pain, such as colitis, appendicitis, irritable bowel syndrome, cholelithiasis, interstitial cystitis, cystitis, urolithiasis, and other conditions that, according to the investigator's judgement, are not suitable for the trial
7. Known or suspected gynecological complaints e.g., premenstrual abdominal pain, deep dyspareunia, uterine fibroids and polyps, or chronic pain (abdominal, dorsal, urogenital)
8. Known instable diseases e.g., psychiatric, cardiovascular, or endocrine disorders
9. Body mass index <18.5 or >34.9 kg/m² at Screening
10. Known or suspected acute infection of gonorrhea, syphilis and/or chlamydia at Screening
11. Current or past estrogen sensitive cancer or pituitary disorder that, in the investigator's opinion, would make the patient not suitable for the trial
12. Women who are breastfeeding, pregnant (positive pregnancy test at Screening), or planning to become pregnant during the trial
13. Fewer than 3 menstrual cycles before Screening following delivery, abortion, miscarriage, or lactation
14. Current severe physical or mental illness
15. Patient does not agree to avoid daily smoking
16. History of alcohol, drug, or medicine abuse within 1 year prior to Screening, or positive for drugs or medicines of abuse in the laboratory analysis performed at Screening
17. Patients with hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption
18. Hypersensitivity to Vitex agnus-castus, lactose or any of the excipients of the IMP or to any ingredients of the standard pain relief medication
19. Patients committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
20. Employees of the sponsor or site staff or direct relatives of the site staff
21. Legal incapacity or limited legal capacity
22. Patients not able to follow trial instructions or assessments or to participate in the trial for the whole duration of approximately 7 months or unable to understand written and verbal instruction, in particular regarding the risks and inconveniences that the patients will be exposed to during participation in the clinical trial
23. Participation in another interventional clinical trial during the last month before Screening
24. Use of Vitex agnus-castus containing preparation or product within the last 3 months before Screening
25. Current intake or intake within the last 4 weeks before Screening of dopamine agonists, dopamine antagonists, estrogens, or antiestrogens that would make the patient not suitable for the trial

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 335 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who respond to treatment defined as: a) a ≥3-point reduction in the peak pelvic pain score and b) no increase in the number of standard pain relief medication | Change from Baseline (28 days prior to randomization) to the cramping window of Cycle No. 5 (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  Response to treatment will be determined by comparing the peak pelvic pain score (using an 11-point numeric rating scale (NRS, scale ranging from 0 (no symptom) to 10 (extreme severity of symptom) of the dysmenorrhea daily diary (DysDD) assessments) made during the cramping window of Cycle 5 with those made at Baseline and by comparing the assessments of number of tablets or capsules of standard pain relief medication taken during the cramping window of Cycle 5 with those taken at Baseline.

SECONDARY OUTCOMES:
Proportion of patients who respond to treatment defined as: a) a ≥3-point reduction in the peak pelvic pain score and b) no increase in the number of standard pain relief medication in the cramping window of Cycles 3, 4, and 6 compared to Baseline | Change from Baseline (28 days prior to randomization) to the cramping windows of Cycles No. 3, 4 and 6 (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  Response to treatment will be determined by comparing the peak pelvic pain score (using an 11-point numeric rating scale (NRS, scale ranging from 0 (no symptom) to 10 (extreme severity of symptom) of the dysmenorrhea daily diary (DysDD) assessments) made during the cramping window of Cycles No. 3, 4 and 6 with those made at Baseline and by comparing the assessments of number of tablets or capsules of standard pain relief medication taken during the cramping window of Cycles No. 3, 4 and 6 with those taken at Baseline.
Proportion of patients with a ≥3-point reduction in the peak pelvic pain score and a decrease in the number of standard pain relief medication | Change from Baseline (28 days prior to randomization) to the cramping windows of Cycles No. 3, 4, 5 and 6) (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The ≥3-point reduction in the peak pelvic pain score using an 11-point numeric rating scale (NRS; scale ranging from 0 (no symptom) to 10 (extreme severity of symptom)) of the dysmenorrhea daily diary (DysDD) will be assessed and the amount of standard pain relief medication taken will be evaluated to investigate the efficacy of the study drug.
Proportion of patients with a peak pelvic pain score of "0" or "1" and no use of standard pain relief medication | At the cramping windows of Cycles No. 3, 4, 5 and 6) (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  Peak pelvic pain score of "0" or "1" using an 11-point numeric rating scale (NRS; scale ranging from 0 (no symptom) to 10 (extreme severity of symptom)) of the dysmenorrhea daily diary (DysDD) and no use of standard pain relief medication during the cramping window of Cycles 3, 4, 5, and 6 will be evaluated.
Assessment of change of peak pelvic pain score | Change from Baseline (28 days prior to randomization) to the cramping windows of Cycles No. 3, 4, 5 and 6) (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The peak pelvic pain score will be assessed using an 11-point numeric rating scale (NRS, scale ranging from 0 (no symptom) to 10 (extreme severity of symptom)) of the dysmenorrhea daily diary (DysDD) assessments and compared to Baseline.
Assessment of the sum of the pelvic pain scores | At the cramping windows of Cycles No. 3, 4 and 5 (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The pelvic pain scores assessed during the cramping windows (4 days) of Cycles 3, 4, and 5 (i.e., 12 assessments in total) using an 11-point numeric rating scale (NRS; scale ranging from 0 (no symptom) to 10 (extreme severity of symptom)) of the dysmenorrhea daily diary (DysDD) will be summed up.
Assessment of the change of the sum of the pelvic pain scores | Change from Baseline (28 days prior to randomization) to the cramping windows of Cycles No. 3, 4, 5 and 6) (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The pelvic pain scores assessed during the cramping window using an 11-point numeric rating scale (NRS, scale ranging from 0 (no symptom) to 10 (extreme severity of symptom)) of the dysmenorrhea daily diary (DysDD) assessments will be summed up per cycle and compared to Baseline.
Assessment of the change in the number of days with pelvic pain | Change from Baseline (28 days prior to randomization) to the cramping windows of Cycles No. 3, 4, 5 and 6) (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The number of days with pelvic pain will be calculated as sum of the days with a pelvic pain above 0 on the 11-point numeric rating scale (NRS, scale ranging from 0 (no symptom) to 10 (extreme severity of symptom)) during the respective cramping window and compared to Baseline.
Assessment of change in the number of standard pain relief medication taken | Change from Baseline (28 days prior to randomization) to the cramping windows of Cycles No. 3, 4, 5 and 6) (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The number of standard pain relief medication will be calculated as sum of the tablets/capsules taken during the respective cramping window and compared to Baseline.
Assessment of change in the number of days with use of standard pain relief medication | Change from Baseline (28 days prior to randomization) to the cramping windows of Cycles No. 3, 4, 5 and 6) (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The number of days with use of standard pain relief medication will be calculated as sum of days with intake of standard pain relief medication during the respective cramping window and compared to Baseline.
Proportion of patients with no use of standard pain relief medication | At the cramping window of Cycle No. 6 (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The number of patients who did not use any standard pain relief medication will be determined.
  The analysis will be performed for all patients as well as for the subgroup of patients who took any standard pain relief medication during the cramping window of Cycle 5.
Assessment of change in the impact on the patient's daily life | Change from Baseline (28 days prior to randomization) to the cramping windows of Cycles No. 3, 4, 5 and 6) (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The impact of pelvic pain or cramps on the patient's daily life including paid work, work around the home, or school work will be assessed on a 5-point scale being part of the dysmenorrhea daily diary (DysDD) assessments (0=not at all, 1=slightly, 2=moderately, 3=quite a bit, 4=extremely). The assessments made during each cramping window will be summed up.
  The impact on physical activities, social or leisure activities, and sleep will be analyzed analogously. The missed time of paid work, work around the home, or school work will be summed up for the cramping window and tabulated by treatment group and cycle.
Investigator's and patient's overall assessment of efficacy using a 5-point verbal rating scale | Visits 4 (Day 85) and 5 (Day 113)
  The treatment efficacy will be assessed by the investigator and the patient using a 5-point verbal rating scale with the following 5 categories: very good, good, moderate, poor, very poor.
Assessment of change in the intensity of menstrual bleeding | Change from Baseline (28 days prior to randomization) to the cramping windows of Cycles No. 3, 4, 5 and 6) (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The intensity of the menstrual bleeding will be assessed on a 5-point scale (0=no bleeding, 1=very light bleeding or spotting, 2=light bleeding, 3=moderate bleeding, 4=heavy bleeding). The assessments made during each cramping window will be summed up.
Assessment of change in the number of pieces of sanitary protection used | Change from Baseline (28 days prior to randomization) to the cramping windows of Cycles No. 3, 4, 5 and 6) (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The number of pieces of sanitary protection used will be assessed on a 4-point scale (0=0, 1=1 piece, 2=2 pieces, 3=3 or more pieces). The assessments made during Day 1 to Day 3 of the cramping window will be summed up.
Assessment of change in the severity of nausea, vomiting, diarrhea, fatigue, weakness, fainting, and headache on a numeric rating scale (NRS) | Change from Baseline (28 days prior to randomization) to the Days 1-3 of Cycles No. 3, 4, 5 and 6 (each cycle is 28 days).
  The analysis is based on the peak NRS score of days 1, 2, and 3 per cycle (11-point NRS scale ranging from 0 (no symptom) to 10 (extreme severity of symptom)).
Proportion of patients with migraine | At Baseline (28 days prior to randomization) and Visits 0, 1, 2, 3, 4 and 5 (i.e., Days 1, 29, 57, 85, 113 and 141)
  The number of patients with migraine will be determined. The chance of patients having a migraine episode since the last clinical trial visit will be analyzed.
Assessment of change in the peak pelvic pain score | At the cramping windows of Cycles No. 5 and 6 (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The change in peak pelvic pain score using an 11-point numeric rating scale (NRS, scale ranging from 0 (no symptom) to 10 (extreme severity of symptom) of the dysmenorrhea daily diary (DysDD) assessments) from cramping window of Cycle 5 to cramping window of Cycle 6 will be analyzed.
Assessment of relative change in the peak pelvic pain score | At the cramping window of Cycles No. 5 and 6 (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The relative change in peak pelvic pain score using an 11-point numeric rating scale (NRS, scale ranging from 0 (no symptom) to 10 (extreme severity of symptom) of the dysmenorrhea daily diary (DysDD) assessments) from cramping window of Cycle 5 to cramping window of Cycle 6 will be analyzed.
Assessment of change in the number of standard pain relief medication taken | At the cramping window of Cycles No. 5 and 6 (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The number of standard pain relief medication will be calculated as sum of tablets/capsules taken during the cramping window. The change from cramping window of Cycle 5 to cramping window of Cycle 6 will be analyzed.
Assessment of relative change in the number of standard pain relief medication taken | At the cramping window of Cycles No. 5 and 6 (each cycle is 28 days). The cramping window is defined as Days -1 to 3 of a menstrual cycle (i.e., 4 days in total).
  The number of standard pain relief medication will be calculated as sum of tablets/capsules taken during the cramping window. The relative change from cramping window of Cycle 5 to cramping window of Cycle 6 will be analyzed.

OTHER OUTCOMES:
Proportion of patients with treatment-emergent adverse events (TEAEs), TEAEs related to the IMP, serious TEAEs related to the IMP, and TEAEs leading to premature discontinuation of the IMP | From Baseline (28 days prior to randomization) until Visit 5 (Day 141).
  The number of patients with TEAEs, TEAEs related to the IMP, serious TEAEs related to the IMP and TEAEs leading to premature discontinuation of the IMP will be determined.
Assessment of change in safety laboratory parameters analyzed from blood samples (hematology) | Change from Baseline (28 days prior to randomization) to Visit 4 (Day 113).
  Proportion of participants with changes in hematology safety laboratory test results will be assessed. Hematology safety parameters which will be analyzed from patients' blood samples include:
  Platelets, hemoglobin, hematocrit, white blood cell count total and differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), red blood cell count, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC).
Assessment of change in safety laboratory parameters analyzed from blood samples (biochemistry) | Change from Baseline to (28 days prior to randomization) Visit 4 (Day 113).
  Proportion of participants with changes in safety laboratory test results will be assessed. Biochemistry safety parameters which will be analyzed from patients' blood samples include:
  Liver: aspartate aminotransferase, alanine aminotransferase, gammaglutamyl transferase, alkaline phosphatase, bilirubin total; Kidney: urea (blood urea nitrogen calculated), creatinine, uric acid, glomerular filtration rate (Cockcroft and Modification of Diet in Renal Disease [MDRD] or Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation), creatine clearance (Cockcroft-Gault) Other: total protein, potassium, sodium, calcium, creatine phosphokinase, glucose, chloride, inorganic phosphorous, lactate dehydrogenase, triglycerides, cholesterol total, albumin.
Assessment of change in vital signs: systolic and diastolic blood pressure | Change from Baseline (28 days prior to randomization) to Visit 4 (Day 113).
  Number of participants with changes in systolic and diastolic blood pressure will be assessed.
Assessment of change in vital signs: pulse | Change from Baseline to (28 days prior to randomization) Visit 4 (Day 113).
  Number of participants with changes in pulse will be assessed.
Assessment of change in vital signs: body temperature | Change from Baseline to (28 days prior to randomization) Visit 4 (Day 113).
  Number of participants with changes in body temperature will be assessed.
Assessment of change in vital signs: body height | Change from Baseline to (28 days prior to randomization) Visit 4 (Day 113).
  Number of participants with changes in body height will be assessed.
Assessment of change in vital signs: body weight | Change from Baseline to (28 days prior to randomization) Visit 4 (Day 113).
  Number of participants with changes in body weight will be assessed.
Assessment of change in physical examination of the genitourinary system: speculum examination | Change from Baseline (28 days prior to randomization) to Visit 4 (Day 113).
  Number of participants with changes in speculum examination findings will be assessed.
Assessment of change in physical examination of the genitourinary system: bimanual examination | Change from Baseline (28 days prior to randomization) to Visit 4 (Day 113).
  Number of participants with changes in bimanual examination findings will be assessed.
Assessment of change in physical examination: palpation of the breast | Change from Baseline (28 days prior to randomization) to Visit 4 (Day 113).
  Number of participants with changes in palpation of the breast findings will be assessed.
Assessment of investigator's and patient's tolerability using a 5-point verbal rating scale | Visits 4 (Day 113) and 5 (Day 141).
  The tolerability will be assessed by investigator and patient using a 5-point verbal rating scale: Very good = 0 (no side effects; no limitation of work and leisure activities due to side effects or adverse reactions); Good = 1 (hardly any side effects; hardly any limitation of work and leisure activities due to side effects or adverse reactions); Moderate = 2 (mild side effects; slight limitation of work and leisure activities due to side effects or adverse reactions); Poor = 3 (distinct side effects; distinct limitation of work and leisure activities due to side effects or adverse reactions); Very poor = 4 (severe side effects; work and leisure activities not possible due to side effects or adverse reactions).
Number of participants with absolute and relative changes in blood hormone concentrations | Changes from Baseline (28 days prior to randomization) to the Visits 2 (Day 57), 3 (Day 85) and 4 (Day 113).
  Absolute and relative changes from Baseline in blood hormone concentration will be analyzed using laboratory tests.
Assessment of change in blood cytokine concentrations | Change from Baseline (28 days prior to randomization) to Visit 4 (Day 113).
  Absolute and relative changes from Baseline in cytokine concentration will be analyzed using Enzyme-linked Immunosorbent Assays (ELISA).
Assessment of change in metabolome parameters (only for optional sub-study) | Change from Baseline (28 days prior to randomization) to Visit 4 (Day 113).
  Absolute and relative changes from Baseline in metabolome parameters assessed in the optional sub-study will be analyzed.
Assessment of change in lipidome parameters (only for optional sub-study) | Change from Baseline (28 days prior to randomization) to Visit 4 (Day 113).
  Absolute and relative changes from Baseline in lipidome parameters assessed in the optional sub-study will be analyzed.
Assessment of change in microbiome parameters (only for optional sub-study) | Change from Baseline (28 days prior to randomization) to Visit 4 (Day 113).
  Absolute and relative changes from Baseline in microbiome parameters assessed in the optional sub-study will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Stute, Prof. Dr., Principal Investigator — Universitätsklinik für Frauenheilkunde, Inselspital Bern
Locations (34):
- Austria (2):
  - Medizinische Universität Innsbruck, Department Frauenheilkunde, Universitätsklinik für Gynäkologische Endokrinologie und Reproduktionsmedizin, Innsbruck
  - Medizinische Universität Wien, Universitätsklinik für Frauenheilkunde, Klinische Abteilung für Gynäkologische Endokrinologie und Reproduktionsmedizin, Vienna
- Czechia (7):
  - Centrum ambulantní gynekologie a primární péče s.r.o., Brno-střed
  - Fakultní nemocnice Brno, Gynekologickoporodnická Klinika, Centrum asistované reprodukce CAR 01 Brno, Brno-střed
  - GYNEKOLOGIE CHEB s.r.o., Cheb
  - NEUMED gynekologická ambulance s.r.o, Olomouc
  - MUDr. Martina Marešová Rosenbergová s.r.o., Pilsen
  - Centrum gynekologické rehabilitace s.r.o, Písek
  - Gyncare MUDr. Michael Švec s.r.o., Plzeň 2-Slovany
- Germany (12):
  - Praxis Dr. Noel, Aachen
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Frauenarztpraxis Dipl. med. Andrea Heweker, Praxis für Gynäkologie, Bernburg
  - Klinische Forschung Dresden GmbH, Dresden
  - Praxis Geseke, Geseke
  - Frauenarztpraxis Dr. Inka Kiesche, Halle
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Frauenarzt-Praxis Dr. med. Klaus Peters, Hamburg
  - Klinische Forschung Hannover Mitte GmbH, Hanover
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Frauenarzt in Stolberg - Wolfgang Clemens, Stolberg
- Hungary (6):
  - Clinexpert Kft., Budapest
  - Óbudai Egészségügyi Centrum Kft., Budapest
  - Zatik Med Kft., Debrecen
  - BKS Research Kft., Hatvan
  - AXON Kereskedelmi Es Szolgaltato Kft., Kecskemét
  - IPR Hungary Kft., Miskolc
- Poland (5):
  - Centrum Medyczne Mikołowska dr Adam Sipiński, Katowice
  - Silmedic Sp. z o.o., Katowice
  - Nzoz Profi-Med, Lublin
  - Centrum Badawcze Panaceum Agnieszka Brzezicka, Magdalena Lenkiewicz Sp. z o.o., Malbork
  - Państwowy Instytut Medyczny Ministerstwa Spraw Wewnętrznych i Administracji, Klinika Położnictwa, Chorób Kobiecych i Ginekologii Onkologicznej, Warsaw
- Sweden (2):
  - Karolinska University Hospital, WHO-centre, Stockholm
  - Umeå University, Dep. of Clinical Sciences, Obstetrics and Gynecology, Umeå